CLINICAL TRIAL: NCT03785964
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 3 Trial of Nirogacestat Versus Placebo in Adult Patients With Progressing Desmoid Tumors/Aggressive Fibromatosis (DT/AF)
Brief Title: Nirogacestat for Adults With Desmoid Tumor/Aggressive Fibromatosis (DT/AF)
Acronym: DeFi
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SpringWorks Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIR-DT-301
Expanded Access: NCT05041036 (Available)
Record Dates: First submitted 2018-12-17; First posted 2018-12-24 (Actual); Results first posted 2024-06-12 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Desmoid Tumor; Aggressive Fibromatosis
Keywords: PF-03084014; GSI; gamma secretase inhibitor; notch pathway
MeSH Terms: conditions — Desmoid Tumors | interventions — nirogacestat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: For the double-blind phase, the participant, investigator, and all other clinical site personnel will be blinded to the assigned treatment allocation. All sponsor personnel will also be blinded except for the sponsor's quality assurance designee(s), safety designee(s), and clinical supply material designee(s).
  Once participants are eligible, they will roll into the open-label phase where they will receive nirogacestat. In the open-label phase, the participant, investigator, all other clinical site personnel, and the sponsor are not blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Double-Blind Phase - Nirogacestat (Experimental): Nirogacestat 150 mg by mouth, twice daily
  Interventions: Drug: Nirogacestat oral tablet
- Double-Blind Phase - Placebo (Placebo Comparator): Placebo by mouth, twice daily
  Interventions: Drug: Placebo Oral Tablet
- Open-Label Phase - Nirogacestat (Experimental): Nirogacestat 150 mg by mouth, twice daily
  Interventions: Drug: Nirogacestat oral tablet

INTERVENTIONS:
Drug: Nirogacestat oral tablet — Nirogacestat tablet
  Other Names: PF-03084014
  Arms: Double-Blind Phase - Nirogacestat; Open-Label Phase - Nirogacestat
Drug: Placebo Oral Tablet — Sugar pill manufactured to mimic nirogacestat 50 mg tablet
  Arms: Double-Blind Phase - Placebo

SUMMARY:
This study evaluates nirogacestat (PF-03084014) in the treatment of desmoid tumor/aggressive fibromatosis (DT/AF). In the double-blind phase, half of the participants will receive nirogacestat while the other half will receive placebo. Once participants are eligible to roll into the open-label phase, they will receive nirogacestat.

DETAILED DESCRIPTION:
Desmoid tumors, also referred to as aggressive fibromatosis, are rare, locally invasive, slow growing soft tissue tumors. Although considered benign because of their inability to metastasize, desmoid tumors can cause significant morbidity and occasionally mortality in patients.

Nirogacestat (PF-03084014) is a potent, small molecule, selective, reversible, noncompetitive inhibitor of γ-secretase (GS) with a potential antitumor activity.

Nirogacestat is being investigated for the treatment of desmoid tumors due to its ability to bind to GS, blocking proteolytic activation of Notch receptors. Previous clinical study data have shown that Notch signaling plays an important role in cancer development. Hence, inhibition of Notch signaling is an important strategy for therapeutic treatment.

ELIGIBILITY:
Double-Blind Key Inclusion Criteria:

* Participant has histologically confirmed DT/AF (by local pathologist prior to informed consent) that has progressed by ≥ 20% as measured by RECIST v1.1 within 12 months of the screening visit scan.
* Participant has:

  1. Treatment naïve, measurably progressing DT/AF that is deemed not amenable to surgery without the risk of significant morbidity; OR
  2. Recurrent, measurably progressing DT/AF following at least one line of therapy; OR
  3. Refractory, measurably progressing DT/AF following at least one line of therapy.
* Participant has a DT/AF tumor where continued progressive disease will not result in immediate significant risk to the participant.
* Participant agrees to provide archival or new tumor tissue for re-confirmation of disease.
* If participant is currently being treated with any therapy for the treatment of DT/AF, this must be completed at least 28 days (or 5 half-lives, whichever is longer) prior to first dose of study treatment. All toxicities from prior therapy must be resolved to ≤Grade 1 or clinical baseline.
* Participants who are receiving chronic nonsteroidal anti-inflammatory drugs (NSAIDs) as treatment for conditions other than DT/AF must be receiving them prior to the documented DT/AF progressive disease (inclusion criteria 2) and on a stable dose for at least 28 days prior to first dose of study treatment.
* Participant has an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 at screening.
* Participant has adequate organ and bone marrow function.

Double-Blind Key Exclusion Criteria:

* Participant has known malabsorption syndrome or preexisting gastrointestinal conditions that may impair absorption of nirogacestat.
* Participant has experienced any of the following within 6 months of signing informed consent: clinically significant cardiac disease (New York Heart Association Class III or IV), myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident, transient ischemic attack, or symptomatic pulmonary embolism.
* Participant has an abnormal QT interval at screening.
* Participant is using concomitant medications that are known to prolong the QT/QTcF interval including Class Ia and Class III antiarrhythmics at the time of informed consent. Non-antiarrhythmic medications which may prolong the QT/QTcF interval are allowed provided the participant does not have additional risk factors for Torsades de Pointes (TdP)
* Participant has congenital long QT syndrome.
* Participant has a history of additional risk factors for Torsades de Pointes (TdP) (e.g., heart failure, hypokalemia, family history of Long QT Syndrome).
* Participant has had lymphoma, leukemia, or any malignancy within the past 5 years at the time of informed consent, except for any locally recurring cancer that has been treated curatively (e.g., resected basal or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of the cervix or breast), with no evidence of metastatic disease for 3 years at the time of informed consent.
* Participant has current or chronic history of liver disease or known hepatic or biliary abnormalities (except for Gilbert's syndrome or asymptomatic gallstones).
* Participant previously received or is currently receiving therapy with GS inhibitors or anti-Notch antibody therapy.
* Participant is currently using any treatment for DT/AF including tyrosine kinase inhibitors (TKIs), NSAIDs (chronic daily use) or any investigational treatment 28 days (or 5 half-lives, whichever is longer) prior to the first dose of study treatment.

OR

Participant has started any treatment for DT/AF after the documented DT/AF progressive disease.

* Participant is currently using or anticipates using food or drugs that are known strong/moderate cytochrome P450 3A4 (CYP3A4) inhibitors, or strong CYP3A inducers within 14 days prior to the first dose of study treatment.
* Participant has a positive human immunodeficiency virus antibody test.
* Participant has presence of Hepatitis B surface antigen at screening.
* Participant has a positive Hepatitis C antibody or Hepatitis C ribonucleic acid (RNA) test result at screening or within 3 months prior to starting study treatment.
* Participant is unable to tolerate MRI or for whom MRI is contraindicated.
* Participant with active or chronic infection at the time of informed consent and during the screening period.
* Participant has experienced other severe acute or chronic medical or psychiatric conditions within 1 year of signing informed consent.
* Participant is unable to comply with study related procedures (including, but not limited to, the completion of electronic patient report outcomes (ePROs), or the ePRO questionnaires are not available in the participant's preferred language).

Open-Label Key Inclusion

* Participant is enrolled in the double-blind phase when the estimated number of PFS events have been observed and the primary PFS analysis has been completed; OR
* Participant is randomized to receive placebo in the double-blind phase and Central Imaging Review determines that the participant has radiographic progressive disease; OR
* Participant is randomized to receive nirogacestat in the double-blind phase and Central Imaging Review determines that the participant has radiographic progressive disease but the participant is deriving clinical benefit without significant toxicity (as determined by the investigator).
* Participant has adequate organ and bone marrow function

Open-Label Key Exclusion

* Participant requires surgery to prevent organ dysfunction.
* Participant has prematurely discontinued from the double-blind phase for any reason other than radiographic progressive disease (as determined by Central Imaging Review).
* Participant developed a concurrent illness/condition that, in the opinion of the investigator, would represent a risk to overall health if they enroll in this study.
* Participant has initiated a new treatment for DT/AF after the Central Imaging Review determines that a participant has radiographic progressive disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2019-04-17 (Actual); Primary Completion 2022-04-07 (Actual); Study Completion 2024-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernd Kasper, MD, Principal Investigator — Mannheim University Medical Center
Locations (52):
- United States (34):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Ronald Regan UCLA Medical Center, Los Angeles, California
  - Stanford Cancer Center, Palo Alto, California
  - UCSF Mission Bay, San Francisco, California
  - Sarcoma Oncology Research Center, Santa Monica, California
  - University of Colorado Hospital-Anschutz Cancer Pavilion (ACP), Aurora, Colorado
  - Smilow Cancer Hospital at Yale-New Haven, New Haven, Connecticut
  - Washington Cancer Institute at MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Mayo Clinic Florida, Jacksonville, Florida
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hosptial (MGH), Boston, Massachusetts
  - Dana-Farber Cancer Institute (DFCI), Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Northwell Health, Lake Success, New York
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - DUMC/Duke Cancer Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - James Cancer Hospital and Solove Research Institute at The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Oregon Health & Science University-Center for Health & Healing, Portland, Oregon
  - Abramson Cancer Center at Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Henry-Joyce Cancer Clinic, Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Wisconsin Clinical Science Center, Madison, Wisconsin
  - Froedtert Hospital & the Medical College of Wisconsin, Milwaukee, Wisconsin
- Belgium (4):
  - Institut Jules Bordet-Medical Oncology, Brussels
  - Cliniques Universitaires Saint-Luc, Institut Roi Albert II, Brussels
  - UZ Gent, Ghent
  - UZ Leuven, Leuven
- Canada (2):
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec
- Germany (3):
  - Helios Klinikum Berlin-Buch, Berlin
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - Universitätsmedizin Mannheim, Mannheim
- Italy (4):
  - IRCCS Istituto Ortopedico Rizzoli, Bologna
  - Istituto di Candiolo IRCCS Oncologia Medica, Candiolo
  - Fondazione IRCCS Instituto Nazionale dei Tumori di Milano, Milan
  - Policlinico Unvrsitario Campus Bio-Medico, Roma
- Netherlands (3):
  - Radboud University Medical Centre, Nijmegen, Gelderland
  - The Netherlands Cancer Institute, Amsterdam
  - Leiden University Medical Center (LUMC), Leiden
- United Kingdom (2):
  - Department of Oncology, University College of London Hospital, London
  - The Royal Marsden NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: Yes
SpringWorks Therapeutics is committed to data transparency and sharing data to further research while maintaining the privacy and confidentiality of research participants. Pertinent patient-level data from completed registrational clinical trials will be made available by SpringWorks to qualified researchers upon approval of reasonable requests following de-identification/anonymization pursuant to applicable law.

REFERENCES:
- [Derived] Ratan R, Kasper B, Alcindor T, Schoffski P, van der Graaf WTA, Federman N, Bui NQ, D'Amato G, Riedel RF, Attia S, Chawla S, Lim A, Tumminello B, Oton AB, Chu Y, Zhou S, Gounder M. Efficacy and Safety of Long-Term Continuous Nirogacestat Treatment in Adults With Desmoid Tumors: Results From the DeFi Trial. J Clin Oncol. 2025 Dec;43(34):3646-3651. doi: 10.1200/JCO-25-00582. Epub 2025 Oct 20. PMID 41115259
- [Derived] Gounder MM, Atkinson TM, Bell T, Daskalopoulou C, Griffiths P, Martindale M, Smith LM, Lim A. GOunder/Desmoid Tumor Research Foundation DEsmoid Symptom/Impact Scale (GODDESS(c)): psychometric properties and clinically meaningful thresholds as assessed in the Phase 3 DeFi randomized controlled clinical trial. Qual Life Res. 2023 Oct;32(10):2861-2873. doi: 10.1007/s11136-023-03445-7. Epub 2023 Jun 22. PMID 37347393
- [Derived] Gounder M, Ratan R, Alcindor T, Schoffski P, van der Graaf WT, Wilky BA, Riedel RF, Lim A, Smith LM, Moody S, Attia S, Chawla S, D'Amato G, Federman N, Merriam P, Van Tine BA, Vincenzi B, Benson C, Bui NQ, Chugh R, Tinoco G, Charlson J, Dileo P, Hartner L, Lapeire L, Mazzeo F, Palmerini E, Reichardt P, Stacchiotti S, Bailey HH, Burgess MA, Cote GM, Davis LE, Deshpande H, Gelderblom H, Grignani G, Loggers E, Philip T, Pressey JG, Kummar S, Kasper B. Nirogacestat, a gamma-Secretase Inhibitor for Desmoid Tumors. N Engl J Med. 2023 Mar 9;388(10):898-912. doi: 10.1056/NEJMoa2210140. PMID 36884323

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Double-Blind Phase - Nirogacestat | Double-Blind Phase - Placebo
Started | 70 | 72
Treated (Safety Population) | 69 | 72
Completed (Completed participants met the study endpoint. Information for completed and not completed pertains to treatment status at the time of the primary analysis. The open-label extension is ongoing.) | 12 | 35
Not Completed | 58 | 37
Not completed — Adverse Event | 14 | 1
Not completed — Unqualified Clinical Progression | 1 | 1
Not completed — Participant non-compliance | 1 | 1
Not completed — Not treated | 1 | 0
Not completed — Other reason | 5 | 11
Not completed — Ongoing (still on treatment) pertains to treatment status at the time of the primary analysis | 36 | 23

BASELINE CHARACTERISTICS:
Population: Intent-To-Treat Population (All Randomized)
Groups:
- Total: Total of all reporting groups
Arm/Group | Double-Blind Phase - Nirogacestat | Double-Blind Phase - Placebo | Total
Number analyzed (Participants) | 70 | 72 | 142
Age, Categorical [Count of Participants; unit: Participants]
  years: <=18 years | 0 | 0 | 0
  years: Between 18 and 65 years | 67 | 69 | 136
  years: >=65 years | 3 | 3 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.5 (14.43) | 37.0 (12.89) | 37.2 (13.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 47 | 92
  Male | 25 | 25 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 9 | 10
  Not Hispanic or Latino | 67 | 55 | 122
  Unknown or Not Reported | 2 | 8 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 5 | 9
  White | 64 | 54 | 118
  More than one race | 1 | 10 | 11
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 4 | 3 | 7
  Netherlands | 4 | 4 | 8
  Belgium | 6 | 5 | 11
  United States | 40 | 50 | 90
  Italy | 5 | 5 | 10
  United Kingdom | 4 | 2 | 6
  Germany | 7 | 3 | 10
Tumor Location (Randomization Stratification Factor) [Count of Participants; unit: Participants] — Count of Participants
  Participants
    Intra-Abdominal | 17 | 18 | 35
    Extra-Abdominal | 53 | 54 | 107

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) Defined as the Time From Randomization Until Date of Assessment of Progression or Death by Any Cause.
Description: Progression will be determined radiographically using RECIST v1.1 (Eisenhauer, 2009) or clinically as assessed by the investigator. Clinical progression is defined as the onset or worsening of symptoms resulting in a global deterioration of health status causing the permanent discontinuation from study treatment and the initiation of emergent treatment (e.g., radiotherapy, surgery, or systemic therapy including chemotherapy or tyrosine kinase inhibitors) for DT/AF. Events of clinical progression will be adjudicated by an independent blinded central Endpoint Adjudication Committee (EAC) which will qualify events of clinical progression for inclusion in the PFS endpoint prior to study unblinding according to an EAC Review Charter.
Time Frame: On the first day of every 3 cycles (each cycle is 28 days) until disease progression is observed or death, whichever comes first, assessed up to approximately 2 years
Population: Intent-to-Treat Population (All Randomized)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Double-Blind Phase - Nirogacestat | Double-Blind Phase - Placebo
Number analyzed (Participants) | 70 | 72
Months | NA [NA to NA] — Not reached. Only less than 50% of the participants had events in Nirogacestat treatment arm. | 15.1 [8.4 to NA] — Upper 95% CI is not reached.
Statistical Analysis 1: Comparison: Double-Blind Phase - Nirogacestat vs Double-Blind Phase - Placebo; Hazard ratio was estimated from stratified Cox proportional hazards model using the exact method for ties, stratified by tumor location. Placebo was the reference treatment; Test type: Superiority; p < 0.001, Log Rank; p-value was from a one-sided stratified log-rank test with placebo as reference; Hazard Ratio (HR) = 0.29, 95% CI 2-sided [0.15 to 0.55]

2. Secondary Outcome: Objective Response Rate Using RECIST Version 1.1 Criteria.
Description: Objective response rate (ORR) is defined as the proportion of participants having a confirmed Best Overall Response (BOR) of CR or PR by central reader using RECIST v1.1 criteria. Responses obtained up until progression, or last evaluable assessment in the absence of progression, will be included in the assessment of ORR. However, any responses, which occurred after a new anticancer therapy was received, will not be included. ORR is presented by percentages of responders.
Time Frame: On the first day of every 3 cycles (each cycle is 28 days) through study completion, an average of 2 years
Population: Intent-to-Treat Population (All Randomized)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Double-Blind Phase - Nirogacestat | Double-Blind Phase - Placebo
Number analyzed (Participants) | 70 | 72
percentage of participants | 41 [29.8 to 53.8] | 8 [3.1 to 17.3]
Statistical Analysis 1: Comparison: Double-Blind Phase - Nirogacestat vs Double-Blind Phase - Placebo; Cochran-Mantel-Haenszel test for general association stratified by tumor location. Placebo was reference treatment; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Two-sided p-value

3. Secondary Outcome: Change From Baseline at Cycle 10 in the Brief Pain Inventory (BPI) Average Pain Intensity (API) Score.
Description: The Brief Pain Inventory consists of 9 questions and utilizes a 11-point Numerical pain Rating Scale from 0-10 measuring severity from "no pain" to "pain as bad as you can imagine," with a 24-hour recall period. Average Pain Intensity is calculated as the 7-day average (when results on at least 4 days for a VISIT are available) of Brief Pain Inventory Question #3 - Worst Pain in last 24 hours. A lower score indicates greater pain relief. The minimum and maximum of the actual score are (0, 8) for Nirogacestat and (0,9) for Placebo, respectively. A positive change from Baseline value indicates worsening of Average Pain Intensity and a negative change from Baseline value indicates improvement of Average Pain Intensity. The minimum and maximum of change from baseline score are (-7, 3) for Nirogacestat and (-5, 5) for Placebo, respectively.
Time Frame: Daily for the last 7 days of every cycle (each cycle is 28 days) through study completion, an average of 2 years
Population: Intent-to-Treat Population
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Double-Blind Phase - Nirogacestat | Double-Blind Phase - Placebo
Number analyzed (Participants) | 70 | 72
score on a scale | -1.583 [-2.157 to -1.009] | -0.241 [-0.822 to 0.340]
Statistical Analysis 1: Comparison: Double-Blind Phase - Nirogacestat vs Double-Blind Phase - Placebo; Mixed model with repeated measures (MMRM) with treatment and visit as factors, Baseline Brief Pain Inventory Short Form score and primary tumor location (intra-abdominal or extra-abdominal) as covariates, included baseline by visit and treatment by visit interactions. Only participants with a Baseline and at least one post-baseline score were included in the analysis. 40 and 31 participants contributed to this analysis at Cycle 10 from Nirogacestat and Placebo respectively; Test type: Superiority; p < 0.001, Mixed Models Analysis; An unstructured covariance structure was used and degrees of freedom were estimated using the Kenward-Roger approximation

4. Secondary Outcome: Change From Baseline at Cycle 10 in the GOunder/Desmoid Tumor Research Tumor Foundation (DTRF) DEsmoid Tumor Symptom Scale (DTSS) - Total Score
Description: The DEsmoid Tumor Symptom Scale is an 11-point, numeric rating scale from 0 to 10 to measure severity from "none" to "as bad as you can imagine," with a 24-hour recall period. The Total Symptom Score is calculated as the mean of Pain items (Items 1-3) as a single score, then a mean of this with items 4-7). Weekly summary scores will be created by averaging the daily scores over the 7 days period prior to each visit. A weekly score will be derived only if 4 or more out of 7 days period have non-missing scores. The weekly summary score will be used in analyses. If no weekly summary score is calculable, the participant will have data considered as missing at that visit. Higher scores represent worse symptom severity. The minimum and maximum of the actual score are (0,7) for Nirogacestat and (0,10) for Placebo. A positive change from Baseline value indicated worsening of symptoms. The minimum and maximum of change from baseline are (-6,1) for Nirogacestat and (-4,5) for Placebo.
Time Frame: Daily for the last 7 days of every cycle (each cycle is 28 days) through study completion, an average of 2 years
Population: Intent-to-Treat Population
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Double-Blind Phase - Nirogacestat | Double-Blind Phase - Placebo
Number analyzed (Participants) | 70 | 72
score on a scale | -1.110 [-1.569 to -0.651] | 0.457 [-0.009 to 0.923]
Statistical Analysis 1: Comparison: Double-Blind Phase - Nirogacestat vs Double-Blind Phase - Placebo; Mixed model with repeated measures (MMRM) with treatment and visit as factors, Baseline DEsmoid Tumor Symptom Scale score and primary tumor location (intra-abdominal or extra-abdominal) as covariates, included baseline by visit and treatment by visit interactions. Only participants with a Baseline and at least one post-baseline score were included in the analysis. 40 and 32 participants contributed to this analysis at Cycle 10 from Nirogacestat and Placebo respectively; Test type: Superiority; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 3, analysis 1]

5. Secondary Outcome: Change From Baseline in the GOunder/Desmoid Tumor Research Foundation (DTRF) DEsmoid Tumor Impact Scale (DTIS) - Physical Functioning Domain Score
Description: The items are evaluated on a 5-point Likert Scale ranging from "none of the time" to "all of the time" to measure frequency, with a 7-day recall period. The Physical Function Domain Score are calculated as the average Item 01 Moving, Item 02 Reaching (Freq), Item 06 Vigorous Activity, Item 7 Moderate Activity, and Item 08 Accomplished Less. Higher scores represent worst impact severity. The minimum and maximum of the actual score are (1, 5) for Nirogacestat and (1,5) for Placebo, respectively. A positive change from baseline value indicates worsening impact and a negative change from baseline value indicates improvement in impact. The minimum and maximum of change from baseline score are (-3, 0) for Nirogacestat and (-1, 2) for Placebo, respectively.
Time Frame: On the last day of every cycle (each cycle is 28 days) through study completion, average of 2 years.
Population: Intent-to-Treat Population
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Double-Blind Phase - Nirogacestat | Double-Blind Phase - Placebo
Number analyzed (Participants) | 70 | 72
score on a scale | -0.613 [-0.808 to -0.418] | 0.094 [-0.113 to 0.300]
Statistical Analysis 1: Comparison: Double-Blind Phase - Nirogacestat vs Double-Blind Phase - Placebo; Mixed model with repeated measures (MMRM) with treatment and visit as factors, Baseline score and primary tumor location (intra-abdominal or extra-abdominal) as covariates, included baseline by visit and treatment by visit interactions. Only participants with a Baseline and at least one post-baseline score were included in the analysis. 39 and 28 participants contributed to this analysis at Cycle 10 from Nirogacestat and Placebo respectively; Test type: Superiority; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 3, analysis 1]

6. Secondary Outcome: Change From Baseline at Cycle10 in the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 (QLQ-C30) Global Health Status/Quality of Life (GHS/QoL) Scale.
Description: The EORTC Quality of Life Questionnaire-Core 30 version 3.0 was used with a 7-day recall period. It consists of 30 questions with all items scored 1 ("not at all") to 4 ("very much") except for the 2 items contributing to the global health status/QoL, which are scored 1 ("very poor") to 7 ("excellent"). The instrument yields the following scales:5 functional scales, 3 symptom scales, and a global health status/quality of life scale. A high score for the global health status/QoL represents a high QoL. The minimum and maximum of the actual score are (33, 100) for Nirogacestat and (8,92) for Placebo, respectively. A positive change from baseline indicated improvement of global health status and a negative change from baseline value indicated worsening of global health status. The minimum and maximum of change from baseline score are (-58, 67) for Nirogacestat and (-67, 42) for Placebo, respectively.
Time Frame: Last day of every cycle (each cycle is 28 days) through study completion, an average of 2 years
Population: Intent-to-Treat Population
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Double-Blind Phase - Nirogacestat | Double-Blind Phase - Placebo
Number analyzed (Participants) | 70 | 72
score on a scale | 2.935 [-3.115 to 8.985] | -8.466 [-15.065 to -1.867]
Statistical Analysis 1: Comparison: Double-Blind Phase - Nirogacestat vs Double-Blind Phase - Placebo; Mixed model with repeated measures (MMRM) with treatment and visit as factors, Baseline score and primary tumor location (intra-abdominal or extra-abdominal) as covariates, included baseline by visit and treatment by visit interactions. Only participants with a Baseline and at least one post-baseline score were included in the analysis. 38 and 27 participants contributed to this analysis at Cycle 10 from Nirogacestat and Placebo respectively; Test type: Superiority; p = 0.006, Mixed Models Analysis; [statistical method as in outcome 3, analysis 1]

7. Secondary Outcome: Change From Baseline at Cycle 10 in the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 (QLQ-C30) Physical Functioning
Description: The EORTC Quality of Life Questionnaire-Core 30 version 3.0 was used with a 7-day recall period. It consists of 30 questions with all items scored 1 ("not at all") to 4 ("very much") except for the 2 items contributing to the global health status/QoL, which are scored 1 ("very poor") to 7 ("excellent"). The instrument yields the following scales:5 functional scales, 3 symptom scales, and a global health status/quality of life scale. A high score for a Physical functional scale represents a high/healthy level of functioning. The minimum and maximum of the actual score are (27, 100) for Nirogacestat and (7,100) for Placebo, respectively. A positive change from baseline indicated improvement of global health status and a negative change from baseline value indicated worsening of physical functioning scores. The minimum and maximum of change from baseline score are (-7, 40) for Nirogacestat and (-40, 27) for Placebo, respectively.
Time Frame: Last day of every cycle (each cycle is 28 days) through study completion, an average of 2 years
Population: Intent-to-Treat Population
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Double-Blind Phase - Nirogacestat | Double-Blind Phase - Placebo
Number analyzed (Participants) | 70 | 72
score on a scale | 9.143 [5.619 to 12.668] | -5.225 [-9.060 to -1.390]
Statistical Analysis 1: Comparison: Double-Blind Phase - Nirogacestat vs Double-Blind Phase - Placebo; Mixed model with repeated measures (MMRM) with treatment and visit as factors, Baseline score and primary tumor location (intra-abdominal or extra-abdominal) as covariates, included baseline by visit and treatment by visit interactions. Only participants with a Baseline and at least one post-baseline score were included in the analysis. 38 and 28 participants contributed to this analysis at Cycle 10 from Nirogacestat and Placebo respectively; Test type: Superiority; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 3, analysis 1]

8. Secondary Outcome: Change From Baseline at Cycle 10 in the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 (QLQ-C30) Role Functioning.
Description: The EORTC Quality of Life Questionnaire-Core 30 version 3.0 was used with a 7-day recall period. It consists of 30 questions with all items scored 1 ("not at all") to 4 ("very much") except for the 2 items contributing to the global health status/QoL, which are scored 1 ("very poor") to 7 ("excellent"). The instrument yields the following scales:5 functional scales, 3 symptom scales, and a global health status/quality of life scale. A positive change from baseline indicated improvement of global health status and a negative change from baseline value indicated worsening of global health status and functioning scores. The minimum and maximum of change from baseline score are (-17, 83) for Nirogacestat and (-100, 50) for Placebo, respectively.
Time Frame: Last day of every cycle (each cycle is 28 days) through study completion, an average of 2 years
Population: Intent-to-Treat Population
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Double-Blind Phase - Nirogacestat | Double-Blind Phase - Placebo
Number analyzed (Participants) | 70 | 72
score on a scale | 13.293 [7.080 to 19.506] | -5.590 [-12.320 to 1.139]
Statistical Analysis 1: Comparison: Double-Blind Phase - Nirogacestat vs Double-Blind Phase - Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 3, analysis 1]

ADVERSE EVENTS:
Time Frame: All SAEs and AEs were collected from the time of signing ICF until 30 days after the last dose of study treatment, an average of 1 years and 4 months and up to 2 years and 10 months. Medical occurrences that begin before the start of study treatment but after obtaining informed consent will be recorded as AEs.
Description: One patient randomized to Nirogacestat arm, discontinued prior to receiving any study drug.
Arm/Group | Double-Blind Phase - Nirogacestat | Double-Blind Phase - Placebo
All-Cause Mortality (participants affected / at risk) | 0/69 | 1/72
Serious Adverse Events (participants affected / at risk) | 14/69 | 8/72
Other Adverse Events (participants affected / at risk) | 69/69 | 69/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-Blind Phase - Nirogacestat (N=69) | Double-Blind Phase - Placebo (N=72)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 2 (2)
Groin abscess (Infections and infestations) | 1 (1) | 0 (0)
Infected cyst (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 3 (4)
Spindle cell sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumor haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Ovarian failure (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Premature menopause (Reproductive system and breast disorders) | 3 (3) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-Blind Phase - Nirogacestat (N=69) | Double-Blind Phase - Placebo (N=72)
Anaemia (Blood and lymphatic system disorders) | 7 (16) | 8 (18)
Abdominal distension (Gastrointestinal disorders) | 4 (4) | 3 (4)
Abdominal pain (Gastrointestinal disorders) | 11 (16) | 9 (18)
Abdominal pain upper (Gastrointestinal disorders) | 5 (6) | 1 (1)
Constipation (Gastrointestinal disorders) | 7 (9) | 7 (8)
Diarrhoea (Gastrointestinal disorders) | 58 (129) | 25 (32)
Dry mouth (Gastrointestinal disorders) | 8 (9) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 6 (6)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 (6) | 3 (3)
Mouth ulceration (Gastrointestinal disorders) | 4 (5) | 0 (0)
Nausea (Gastrointestinal disorders) | 37 (53) | 28 (32)
Stomatitis (Gastrointestinal disorders) | 20 (43) | 3 (3)
Vomiting (Gastrointestinal disorders) | 14 (21) | 14 (17)
Chills (General disorders) | 4 (5) | 1 (1)
Fatigue (General disorders) | 35 (56) | 26 (31)
Influenza like illness (General disorders) | 7 (7) | 2 (2)
Non-cardiac chest pain (General disorders) | 5 (5) | 5 (5)
Oedema peripheral (General disorders) | 4 (5) | 1 (1)
Pyrexia (General disorders) | 5 (7) | 6 (10)
COVID-19 (Infections and infestations) | 12 (12) | 11 (13)
Folliculitis (Infections and infestations) | 9 (25) | 0 (0)
Sinusitis (Infections and infestations) | 6 (9) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 1 (1)
Alanine aminotransferase increased (Investigations) | 12 (17) | 6 (11)
Aspartate aminotransferase increased (Investigations) | 11 (16) | 8 (12)
Blood follicle stimulating hormone increased (Investigations) | 7 (9) | 1 (1)
SARS-CoV-2 test positive (Investigations) | 8 (8) | 10 (10)
Weight decreased (Investigations) | 6 (10) | 7 (8)
Weight increased (Investigations) | 11 (19) | 5 (12)
White blood cell count decreased (Investigations) | 2 (3) | 5 (8)
Decreased appetite (Metabolism and nutrition disorders) | 11 (13) | 8 (11)
Hypokalaemia (Metabolism and nutrition disorders) | 8 (12) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 4 (6) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 29 (66) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (9) | 9 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (10) | 7 (9)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (5)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (6) | 4 (5)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5 (7) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (6) | 6 (6)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 12 (16)
Dizziness (Nervous system disorders) | 8 (10) | 4 (5)
Headache (Nervous system disorders) | 20 (25) | 11 (15)
Memory impairment (Nervous system disorders) | 4 (5) | 2 (2)
Paraesthesia (Nervous system disorders) | 1 (1) | 4 (6)
Anxiety (Psychiatric disorders) | 6 (8) | 5 (6)
Insomnia (Psychiatric disorders) | 6 (11) | 8 (8)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 5 (5) | 0 (0)
Menstruation irregular (Reproductive system and breast disorders) | 6 (6) | 4 (4)
Ovarian failure (Reproductive system and breast disorders) | 12 (14) | 0 (0)
Premature menopause (Reproductive system and breast disorders) | 8 (11) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (18) | 3 (3)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 (15) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7 (11) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 13 (13) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 15 (22) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 11 (13) | 5 (5)
Hidradenitis (Skin and subcutaneous tissue disorders) | 6 (12) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 9 (12) | 6 (6)
Rash (Skin and subcutaneous tissue disorders) | 13 (15) | 5 (6)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 22 (40) | 4 (8)
Hot flush (Vascular disorders) | 13 (14) | 4 (4)
Hypertension (Vascular disorders) | 10 (18) | 8 (11)
Hypotension (Vascular disorders) | 4 (6) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 (5) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol (2021-02-09): https://cdn.clinicaltrials.gov/large-docs/64/NCT03785964/Prot_000.pdf
  • Statistical Analysis Plan: Main SAP (2022-05-12): https://cdn.clinicaltrials.gov/large-docs/64/NCT03785964/SAP_001.pdf
  • Statistical Analysis Plan: Patient-Reported Outcomes (2022-04-05): https://cdn.clinicaltrials.gov/large-docs/64/NCT03785964/SAP_002.pdf